CLINICAL TRIAL: NCT03781323
Title: Neoadjuvant FOLFOX Therapy With Short Course Radiation and Active Surveillance in Locally Advanced Rectal Cancer: A Phase II Study
Brief Title: Neoadjuvant FOLFOX Therapy With Short Course Radiation and Active Surveillance in Locally Advanced Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Richard Dunne, Associate Professor of Hematology/Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGIC18095
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Advanced Rectal Cancer
Keywords: Advanced rectal cancer; FOLFOX (fluorouracil, leucovorin, oxaliplatin)
MeSH Terms: interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin) (Experimental): Patients treated on protocol will be treated with modified FOLFOX. Patients will receive 10 cycles of FOLFOX, administered every other week. FOLFOX will be given on day 1 of each cycle.
  Patients will receive oxaliplatin 85 mg/m² IV over 120 minutes, leucovorin 400 mg/m² IV over 120 minutes, 5-FU 400 mg/m² IVP followed by 5-FU 2400 mg/m² infuse over 46 hours.
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: FOLFOX — Patients treated on protocol will be treated with modified FOLFOX. Patients will receive 10 cycles of FOLFOX, administered every other week. FOLFOX will be given on day 1 of each cycle.
  Patients will receive oxaliplatin 85 mg/m² IV over 120 minutes, leucovorin 400 mg/m² IV over 120 minutes, 5-FU 400 mg/m² IVP followed by 5-FU 2400 mg/m² infuse over 46 hours.

SUMMARY:
The purpose of this study is to evaluate the treatment of patients with locally advanced rectal cancer for complete response to neoadjuvant chemotherapy without the use of radiation and surgery.

DETAILED DESCRIPTION:
These patients will be evaluated for complete clinical response (cCR) after completing 10 cycles of FOLFOX (fluorouracil, leucovorin, oxaliplatin) chemotherapy, with interval analysis after six cycles. Patients who have stable or progressive disease will be treated per discretion of the treating physician following multidisciplinary discussion. Those determined to have partial or complete response will complete full neoadjuvant treatment and undergo close surveillance with watchful waiting for local recurrence without immediate surgery. The primary endpoint of this study will be the rate of cCR, which is to include complete and near complete clinical response, with secondary endpoints of disease free survival (DFS), overall survival (OS), quality of life (QOL), as well as evaluation of safety and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >18 years old at time of diagnosis
2. Histologically confirmed adenocarcinoma of the rectum from biopsy, defined as adenocarcinoma <15 cm from the anal verge
3. Clinical staging including T3N0 tumors, or T1-3 with N1-2a disease
4. Patients with lower rectal cancer deemed by surgery to not be candidates for sphincter sparing surgery are eligible to participate
5. There must be no evidence of metastatic disease any time prior to initiation of study
6. Rectal tumors must be determined as likely requiring total mesorectal excision (TME)
7. Participant must be treatment naïve for rectal cancer, with no prior radiation chemotherapy, radiation, or surgery for specific rectal cancer
8. No history of prior pelvic radiation
9. No prior administration of platinum agents
10. No active infections requiring intravenous antibiotics
11. No additional active malignancy
12. No prior treatment of any malignancy within the past 3 years
13. Baseline lab work must meet the following parameters:

    1. Absolute neutrophil count (ANC)>1500/mm3
    2. Platelet count>100,000/mm3
    3. Hemoglobin>8.0 g/dL
    4. Total bilirubin and creatinine < 1.5x upper limit of normal (ULN)
    5. AST and ALT < 3x ULN
14. Women of childbearing potential (WCBP) will be defined as those biologically capable of becoming pregnant. WCBP must be negative for pregnancy testing (urine or blood) and agree to use effective contraception. Viable contraception should be used after trial screening, before initiation of chemotherapy, and throughout the duration of active treatment in the study.
15. Participants must be read and explained the purposes of the study, and sign a statement of informed consent prior to participation. Those who do not read or understand English are eligible and may be consented according to institutional federal regulations.

Exclusion Criteria:

1. Recurrent or refractory rectal adenocarcinoma
2. T1N0, T2N0, T4a, T4b, or N2b tumors
3. Any evidence of metastatic disease
4. Primary unresectable rectal cancer. A tumor will be considered unresectable when invading adjacent organs such that an en bloc resection cannot achieve negative margins
5. Patients with threatened margins, defined as tumor <1 mm from circumferential resection margins or mesorectal fascia
6. Patients unable to undergo MRI imaging
7. Patient with a history of any arterial thrombotic event within the past 6 months. This includes angina, myocardial infarction, transient ischemic attack, or cerebral vascular accident.
8. Patients with history of venous thrombotic episodes such as deep vein thrombosis, pulmonary embolus occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Patients who are anticoagulated for atrial fibrillation or other conditions may participate only if on stable doses of anticoagulant therapy.
9. Patients with cardiovascular, hepatic, or renal systemic diseases that would preclude use of chemotherapy
10. Peripheral neuropathy>grade 1 by Common Terminology Criteria for Adverse Events, or CTCAEa
11. The patient must not be on any clinical trials involving other experimental therapies before or during study treatment
12. Women who are currently pregnant or breast-feeding
13. Men and women expecting to father/conceive children
14. Patients with any other concord medical or psychiatric condition which were deemed inappropriate for entry into the study per the investigator.
15. History of other invasive malignancy within the past 3 years, except for adequately treated non-melanoma skin cancer, ductal carcinoma in situ, bladder carcinoma in situ or carcinoma in situ of the cervix.

aCTCAE version 5.0 from Department of Health and Human Services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2027-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dunne, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester, James P. Wilmot Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 patients were consented, 1 failed screening
Groups:
- mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin): Patients treated on protocol will be treated with modified FOLFOX. Patients will receive 10 cycles of FOLFOX, administered every other week. FOLFOX will be given on day 1 of each cycle.
  Patients will receive oxaliplatin 85 mg/m² IV over 120 minutes, leucovorin 400 mg/m² IV over 120 minutes, 5-FU 400 mg/m² IVP followed by 5-FU 2400 mg/m² infuse over 46 hours.
  FOLFOX: Patients treated on protocol will be treated with modified FOLFOX. Patients will receive 10 cycles of FOLFOX, administered every other week. FOLFOX will be given on day 1 of each cycle.
  Patients will receive oxaliplatin 85 mg/m² IV over 120 minutes, leucovorin 400 mg/m² IV over 120 minutes, 5-FU 400 mg/m² IVP followed by 5-FU 2400 mg/m² infuse over 46 hours.
Period: Overall Study
Arm/Group | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 51.4 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Complete Clinical Response.
Description: * A complete response will consist of a digital rectal exam with normal appearing mucosa and sigmoidoscopy/proctoscopy with scarring but no nodularity or ulcerations.
  * A near complete response will consist of digital rectal exam with smooth or minor mucosal abnormalities, and sigmoidoscopy/proctoscopy with small mucosal abnormalities, or superficial ulceration or erythematous scarring.
  * Partial response, in our study, will be those tumors read with RECIST version 1.1 criteria with a ≥20% decrease in size without obtaining near or complete response.
  * Stable disease, in our study, will be those tumors read with RECIST criteria with a <20% decrease in size without obtaining near or complete response.
  * Progressive disease will be those tumors with >20% increase in size by RECIST version 1.1 criteria on imaging.
Time Frame: 1 year
Population: Data was missing for one participant.
Measure: Number; unit: proportion or participants
Arm/Group | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin)
Number analyzed (Participants) | 11
proportion or participants | 0.27

2. Secondary Outcome: Proportion of Patients With Survival
Description: Will be measured by physical exams
Time Frame: 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients With Survival
Description: Will be measured by laboratory testing
Time Frame: 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Patients With Survival
Description: Will be measured by proctoscopy
Time Frame: 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Patients With Survival
Description: Will be measured by sigmoidoscopy
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin)
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin) (N=12)
acute kidney injury (Renal and urinary disorders) | 1
Sepsis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
colonic performation (Gastrointestinal disorders) | 1
colitis (Gastrointestinal disorders) | 1
ileus (Gastrointestinal disorders) | 1
ileal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX (5-Fluorouracil Leucovorin Oxaliplatin) (N=12)
abdominal pain (Gastrointestinal disorders) | 5
alanine aminotransferase increase (Investigations) | 1
alkaline phosphatase increased (Investigations) | 1
alopecia (Skin and subcutaneous tissue disorders) | 1
anemia (Blood and lymphatic system disorders) | 3
anorexia (Metabolism and nutrition disorders) | 1
anxiety (Nervous system disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
atrial fibrillation (Cardiac disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
Mediport Thrombus (Blood and lymphatic system disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Edema limbs (General disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Abdominal Cramping (Gastrointestinal disorders) | 1
Hypoactive Bowel Sounds (Gastrointestinal disorders) | 1
Mouth sores (Gastrointestinal disorders) | 1
Cold Sensitivity in hand and throat (General disorders) | 1
Headache (Nervous system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothermia (General disorders) | 1
Mediport Incision Infection (Infections and infestations) | 1
Lesion from tick bite on upper back (Injury, poisoning and procedural complications) | 1
Insomnia (Nervous system disorders) | 2
Lip infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Neck/Jawline pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Cold Sensitivity (Nervous system disorders) | 1
Sleep Disturbance (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (General disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Palpitations (Cardiac disorders) | 2
Paresthesia (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 7
Platelet count decreased (Investigations) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep Disturbance (Psychiatric disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Vaginal spotting (Reproductive system and breast disorders) | 1
Sepsis (Infections and infestations) | 1
Nasal Sores (Skin and subcutaneous tissue disorders) | 1
Irritant dermatitis around stoma (Skin and subcutaneous tissue disorders) | 2
Diaphoretic (Skin and subcutaneous tissue disorders) | 1
Erythema to fingertips (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Wound complication (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT03781323/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT03781323/ICF_001.pdf